CLINICAL TRIAL: NCT03559777
Title: Evaluation for Primary Stability of Implant in Closed Sinus Lifting Cases Using Densah Bur Versus Osteotome in Partially Edentulous Patients (A Randomized Clinical Trial)
Brief Title: Primary Stability of Implant in Closed Sinus Lifting Cases Using Densah Bur Versus Osteotome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Taha amer taha, Principal Investigator(doctor), Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: closed sinus lifiting
Record Dates: First submitted 2018-06-05; First posted 2018-06-18 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Sinus Pneumatization
Keywords: closed sinus lifiting; implant stability; osteotome; densah bur

STUDY DESIGN:
Intervention Model Description: The patients will be randomly divided into 2 equal groups
Who Masked: Investigator
Masking Description: Each patient will be given a code by the researcher and the observers will be blind to which group this case belong.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- closed sinus lifting by Osteotome (Active Comparator): * Local anesthesia will be injected intra-orally
  * A full thickness flap will be elevated
  * A pilot drill will be used to start the osteotomy preparation, which should be ended 1mm short of sinus floor.
  * The widening drills can be sequentially used to widen the osteotomy site to the same level
  * An osteotome of diameter a little less than the planned implant body, will be inserted in the prepared osteotomy site and gently tapped to reach the same level.
  * The osteotome will be tapped gently to fracture up the sinus floor.
  * Xenograft will be added to the osteotomy as the grafting material.
  * Once the desired height of sinus elevation will be gained and grafted, the implant fixture will be inserted.
  * Smart peg will be placed on implant and Ostell will be used to record ISQ.
  * Healing collar will be placed on implant.
  * Suturing the flab around healing collar.
  Interventions: Other: closed sinus lifting by Osteotome
- closed sinus lifting by Densah bur (Experimental): * Local anesthesia will be injected intra-orally
  * A full thickness flap will be elevated
  * A pilot drill will be used to start the osteotomy , which should be ended 1mm short of sinus floor.
  * Change the drill motor to reverse- densifying Mode
  * Begin with the densah bur (2.5mm) until 1 mm short of the sinus floor.
  * Use the next wider Densah Bur (3.0) in densifying-mode until feeling the haptic feedback of the bur reaching the dense sinus floor, modulate pressure with a gentle pumping motion to advance past the sinus floor in 1 mm increments.
  * densah burs (3.5mm) advance in the osteotomy.
  * Xenograft will be added to the osteotomy .
  * Once the desired height of sinus elevation will be gained and grafted, the implant fixture will be inserted.
  * Smart peg will be placed on implant and Ostell will be used to record ISQ.
  * Healing collar will be placed on implant.
  * Suturing the flab around healing collar.
  Interventions: Other: closed sinus lifting by Densah bur

INTERVENTIONS:
Other: closed sinus lifting by Osteotome — * Local anesthesia will be injected intra-orally
  * A full thickness flap will be elevated
  * A pilot drill will be used to start the osteotomy preparation, which should be ended 1mm short of sinus floor.
  * The widening drills can be sequentially used to widen the osteotomy site to the same level
  * An osteotome of diameter a little less than the planned implant body, will be inserted in the prepared osteotomy site and gently tapped to reach the same level.
  * The osteotome will be tapped gently to fracture up the sinus floor.
  * Xenograft will be added to the osteotomy as the grafting material.
  * Once the desired height of sinus elevation will be gained and grafted, the implant fixture will be inserted.
  * Smart peg will be placed on implant and Ostell will be used to record ISQ.
  * Healing collar will be placed on implant.
  * Suturing the flab around healing collar.
  Arms: closed sinus lifting by Osteotome
Other: closed sinus lifting by Densah bur — * Local anesthesia will be injected intra-orally
  * A full thickness flap will be elevated
  * A pilot drill will be used to start the osteotomy , which should be ended 1mm short of sinus floor.
  * Change the drill motor to reverse- densifying Mode
  * with the densah bur (2.5mm) until 1 mm short of the sinus floor.
  * Use the next wider Densah Bur (3.0) in densifying-mode until feeling the haptic feedback of the bur reaching the dense sinus floor, modulate pressure with a gentle pumping motion to advance past the sinus floor in 1 mm increments.
  * densah burs (3.5mm) advance in the osteotomy.
  * Xenograft will be added to the osteotomy .
  * Once the desired height of sinus elevation will be gained and grafted, the implant fixture will be inserted.
  * Smart peg will be placed on implant and Ostell will be used to record ISQ.
  * Healing collar will be placed on implant.
  * Suturing the flab around healing collar.
  Arms: closed sinus lifting by Densah bur

SUMMARY:
This study is aiming to evaluate primary stability of implant in closed sinus lifting cases by Densah bur in compared to Osteotome in partially edentulous patients hoping that densah bur can lift the sinus membrane and improve primary stability of implant.

DETAILED DESCRIPTION:
The osteotome technique is effective in certain cases, but the most sensitive aspect is the tapping force, which should be sufficient enough to infracture the sinus floor cortical bone but restrained enough to prevent the osteotome tip from traumatizing the Schneiderian membrane.

Several surgical techniques have been proposed to minimize the sinus membrane perforation rate by using a piezosurgical device, balloon, hydrostatic pressure.

The success of therapy in posterior maxilla is not only dependent on the success of the sinus elevation but also the primary stability of the implant that allow bone apposition on the implant surface without any micromovement for osseeointegration.

Later, densah burs are introduced as another treatment option for internal transalveolar approach of sinus floor elevation with improving primary stability of implant by osseodensification.

As treatment options of edentulous maxillary today may include dental implants, the practitioner must be familiar with various sinus lift surgical techniques in order to choose an ideal treatment option for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Both males as well as females without any active periodontal disease.
* All patients were in a good health with no systemic diseases.
* All selected patients were non-smokers and non-alcoholics.
* Patient were free from T.M.J troubles, abnormal oral habits such as bruxism.
* The edentulous ridges were covered with optimal thickness of soft tissue.
* Remaining natural teeth had good.
* Periodontal tissue support and occlusion showed sufficient inter arch space.
* On the local level, patients with maxillary sinus diseases and unfavorable inter maxillary relationship were excluded.

Exclusion Criteria:

* Patients with residual bone height less than 6mm.
* Patients with systemic disease that may affect bone quality.
* Patients with poor oral hygiene and active periodontal diseases.
* Patient with limited mouth opening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
stability of implant | Implant stability will be measured intraoperative at time of surgery
  After implant placement, Implant stability will be measured by Ostell
stability of implant | Implant stability will be measured at second week
  Implant stability will be measured by Ostell
stability of implant | Implant stability will be measured at fourth week
  Implant stability will be measured by Ostell
stability of implant | Implant stability will be measured at the sixth week
  Implant stability will be measured by Ostell
stability of implant | Implant stability will be measured at The eighth week
  Implant stability will be measured by Ostell

REFERENCES:
- [Background] Zohrabian VM, Sonick M, Hwang D, Abrahams JJ. Dental Implants. Semin Ultrasound CT MR. 2015 Oct;36(5):415-26. doi: 10.1053/j.sult.2015.09.002. Epub 2015 Sep 12. PMID 26589695
- [Background] Atwood DA. Reduction of residual ridges: a major oral disease entity. J Prosthet Dent. 1971 Sep;26(3):266-79. doi: 10.1016/0022-3913(71)90069-2. No abstract available. PMID 4934947
- [Background] Tatum H Jr. Maxillary and sinus implant reconstructions. Dent Clin North Am. 1986 Apr;30(2):207-29. PMID 3516738
- [Background] Valentini P, Abensur DJ. Maxillary sinus grafting with anorganic bovine bone: a clinical report of long-term results. Int J Oral Maxillofac Implants. 2003 Jul-Aug;18(4):556-60. PMID 12939008
- [Background] Summers RB. A new concept in maxillary implant surgery: the osteotome technique. Compendium. 1994 Feb;15(2):152, 154-6, 158 passim; quiz 162. PMID 8055503
- [Background] Pjetursson BE, Tan WC, Zwahlen M, Lang NP. A systematic review of the success of sinus floor elevation and survival of implants inserted in combination with sinus floor elevation. J Clin Periodontol. 2008 Sep;35(8 Suppl):216-40. doi: 10.1111/j.1600-051X.2008.01272.x. PMID 18724852
- [Background] Chen L, Cha J. An 8-year retrospective study: 1,100 patients receiving 1,557 implants using the minimally invasive hydraulic sinus condensing technique. J Periodontol. 2005 Mar;76(3):482-91. doi: 10.1902/jop.2005.76.3.482. PMID 15857085
- [Background] Pietrokovski J, Massler M. Alveolar ridge resorption following tooth extraction. J Prosthet Dent. 1967 Jan;17(1):21-7. doi: 10.1016/0022-3913(67)90046-7. No abstract available. PMID 5224784
- [Background] Bartee BK. Extraction site reconstruction for alveolar ridge preservation. Part 1: rationale and materials selection. J Oral Implantol. 2001;27(4):187-93. doi: 10.1563/1548-1336(2001)0272.3.CO;2. PMID 12500877
- [Background] Sharan A, Madjar D. Maxillary sinus pneumatization following extractions: a radiographic study. Int J Oral Maxillofac Implants. 2008 Jan-Feb;23(1):48-56. PMID 18416412
- [Background] Chrcanovic BR, Albrektsson T, Wennerberg A. Reasons for failures of oral implants. J Oral Rehabil. 2014 Jun;41(6):443-76. doi: 10.1111/joor.12157. Epub 2014 Mar 11. PMID 24612346
- [Background] Geckili O, Bilhan H, Geckili E, Cilingir A, Mumcu E, Bural C. Evaluation of possible prognostic factors for the success, survival, and failure of dental implants. Implant Dent. 2014 Feb;23(1):44-50. doi: 10.1097/ID.0b013e3182a5d430. PMID 24113554
- [Background] Lundgren S, Cricchio G, Hallman M, Jungner M, Rasmusson L, Sennerby L. Sinus floor elevation procedures to enable implant placement and integration: techniques, biological aspects and clinical outcomes. Periodontol 2000. 2017 Feb;73(1):103-120. doi: 10.1111/prd.12165. PMID 28000271
- [Background] Schwartz-Arad D, Herzberg R, Dolev E. The prevalence of surgical complications of the sinus graft procedure and their impact on implant survival. J Periodontol. 2004 Apr;75(4):511-6. doi: 10.1902/jop.2004.75.4.511. PMID 15152813
- [Background] Tan WC, Lang NP, Zwahlen M, Pjetursson BE. A systematic review of the success of sinus floor elevation and survival of implants inserted in combination with sinus floor elevation. Part II: transalveolar technique. J Clin Periodontol. 2008 Sep;35(8 Suppl):241-54. doi: 10.1111/j.1600-051X.2008.01273.x. PMID 18724853
- [Background] Di Girolamo M, Napolitano B, Arullani CA, Bruno E, Di Girolamo S. Paroxysmal positional vertigo as a complication of osteotome sinus floor elevation. Eur Arch Otorhinolaryngol. 2005 Aug;262(8):631-3. doi: 10.1007/s00405-004-0879-9. Epub 2005 Feb 27. PMID 15735973
- [Background] Garbacea A, Lozada JL, Church CA, Al-Ardah AJ, Seiberling KA, Naylor WP, Chen JW. The incidence of maxillary sinus membrane perforation during endoscopically assessed crestal sinus floor elevation: a pilot study. J Oral Implantol. 2012 Aug;38(4):345-59. doi: 10.1563/AAID-JOI-D-12-00083. PMID 22913307
- [Background] Nobrega AR, Norton A, Silva JA, Silva JP, Branco FM, Anitua E. Osteotome versus conventional drilling technique for implant site preparation: a comparative study in the rabbit. Int J Periodontics Restorative Dent. 2012 Jun;32(3):e109-15. PMID 22408780
- [Background] Buchter A, Kleinheinz J, Wiesmann HP, Kersken J, Nienkemper M, Weyhrother Hv, Joos U, Meyer U. Biological and biomechanical evaluation of bone remodelling and implant stability after using an osteotome technique. Clin Oral Implants Res. 2005 Feb;16(1):1-8. doi: 10.1111/j.1600-0501.2004.01081.x. PMID 15642025
- [Background] Stavropoulos A, Nyengaard JR, Lang NP, Karring T. Immediate loading of single SLA implants: drilling vs. osteotomes for the preparation of the implant site. Clin Oral Implants Res. 2008 Jan;19(1):55-65. doi: 10.1111/j.1600-0501.2007.01422.x. Epub 2007 Oct 22. PMID 17956566
- [Background] Rosen PS, Summers R, Mellado JR, Salkin LM, Shanaman RH, Marks MH, Fugazzotto PA. The bone-added osteotome sinus floor elevation technique: multicenter retrospective report of consecutively treated patients. Int J Oral Maxillofac Implants. 1999 Nov-Dec;14(6):853-8. PMID 10612923
- [Background] Meyer, E, and S Huwais, 'Osseodensification Is a Novel Implant Preparation Technique That Increases Implant Primary Stability by Compaction and Auto-Grafting Bone', American Academy of Periodontology, 2014